CLINICAL TRIAL: NCT03021213
Title: Treating Heart Failure With Enhanced External Counterpulsation (EECP): Prospective, Multi-centric Observational Cohort Study
Brief Title: Treating Heart Failure With Enhanced External Counterpulsation (EECP)
Status: Withdrawn | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Campus Virchow - Klinikum, Charité - University Medicine Berlin, Charite University, Berlin, Germany
Other Study IDs: EECP
Record Dates: First submitted 2016-10-27; First posted 2017-01-13 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Enhanced external counterpulsation (EECP) is an outpatient coronary artery disease (CAD) therapy that involves the cyclical inflation/deflation of cuffs wrapped around the lower extremities. However, the possible benefits of EECP in patients with heart failure (HF) (New York Heart Association [NYHA] classes II to IV) and cardiomyopathy are unclear.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure (NYHA II-IV)

  1. with optimal medical therapy
  2. caused by ischemic or non-ischemic cardiomyopathy
* EECP-Therapy and Treatment in the Cardio Centrum Berlin or Charité - University Medicine Berlin
* Aged 18 to 100 years
* Offered patient information and written informed consent

Exclusion Criteria:

* Participation in another interventional trial
* Acute coronary syndrome < 4 weeks prior to enrollment
* Operation < 4 weeks prior to enrollment
* Stroke < 4 weeks prior to enrollment
* Clinically significant disease with hospitalization
* Aortic valvular heart disease ≥ moderate
* Aortic aneurysm
* clinically relevant severe cardiopulmonal diseases
* Resting RR > 160/90mmHg
* Thrombose, Thrombophlebitis < 8 weeks prior to enrollment
* Peripheral artery occlusive disease ≥ Stadium II
* Acute Heart failure
* Pathological bleeding tendency
* Arrhythmias, which interfere with Triggering of the EECP
* Other diseases, that inhibit EECP-Treatment (e.g. Spinal disc herniation)
* Accommodation in an institution due to an official or judicial order
* Women: pregnancy or lactation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure (NYHA II-IV)
  * with optimal medical therapy
  * arisen from ischemic or non-ischemic cardiomyopathy
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic heart function | A period of 1 year

SECONDARY OUTCOMES:
Ergometric power increase | A period of 1 year
  Ergometric power increase will be measured by individuals' performance in ergometric work load. Scale is Watt.
Subjective health Status - Mental Health Composite Score | A period of 1 year
  Sf-12-questionnaire: value of the Mental Health Composite Score
Subjective health Status - Physical Health Composite Score | A period of 1 year
  Sf-12-questionnaire: value of the Physical Health Composite Score
Organ complications | A period of 1 year
  Relevant laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité - University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No